CLINICAL TRIAL: NCT05040672
Title: Evaluation of Knowledge and Practice About Prostate Cancer in Male Employees of Libbs Pharmaceuticals
Brief Title: Evaluation of Knowledge and Practice About Prostate Cancer in Male Employees
Acronym: LB2008
Status: Completed | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB2008
Record Dates: First submitted 2021-08-30; First posted 2021-09-10 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I: All volunteer male employees of Libbs Pharmaceuticals residing in all Brazilian regions will participate in this research.An online questionnaire will be applied to assess research subjects understanding of prostate cancer and health habits.
  Interventions: Behavioral: questionare online application

INTERVENTIONS:
Behavioral: questionare online application — questionare online application

SUMMARY:
Analyze, through an online questionnaire, the knowledge and practice about the prevention and detection of prostate cancer in male employees of a pharmaceutical company.

DETAILED DESCRIPTION:
In Brazil, there are still few published and current studies that explore man's attention and awareness of health. Historically, women attend medical appointments and perform routine tests more frequently than men. For this is very important Analyze, through an online questionnaire, the knowledge and practice about the prevention and detection of prostate cancer in male employees of Libbs Farmacêutica (a pharmaceutical company in Brazil).

ELIGIBILITY:
Inclusion Criteria:

* Male individuals included in the Libbs workforce;
* Age 18 years or older;
* Subjects who agree to participate in the study after reading and signing the Informed Consent Form.

Exclusion Criteria:

* There is no exclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As this is a non-probabilistic or convenience (non-random) sampling, the sample size calculation is not applicable. Today there are about 1500 male employees at Libbs Pharmaceuticals and all will be invited to participate in the survey. Answers obtained from all questionnaires filled in their entirety will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of Knowledge and Practice About Prostate Cancer e Healthy Habits | 1 month
  Assess the subjects knowledge and practice in relation to educational campaigns aimed at prostate cancer.All the information wil be collected using a questionnaire previously approved by the ethics committee.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Figueiredo, São Paulo, Brazil